CLINICAL TRIAL: NCT06029127
Title: A Phase 2, Open-label, Randomized, Multi-arm Study of BGB-A445 in Combination With Investigational Agents in Non-Small Cell Lung Cancer Patients Previously Treated With Anti-PD-(L)1 Antibody
Brief Title: A Study of Gimistotug (BGB-A445) in Combination With Other Investigational Agents in Participants With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-LC-203; CTR20233070 (Other: ChinaDrugTrials)
Record Dates: First submitted 2023-08-24; First posted 2023-09-08 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: PD-L1; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gimistotug + Docetaxel (Experimental): Participants received gimistotug and docetaxel 75 mg/m^2 both by intravenous infusion once every 3 weeks until disease progression, intolerable toxicity, withdrawal of informed consent, or other discontinuation criterion were met.
  Interventions: Drug: Gimistotug; Drug: Docetaxel
- Gimistotug + BGB-15025 (Experimental): Participants received gimistotug by intravenous infusion once every 3 weeks and BGB-15025 orally once daily during each 3-week cycle until disease progression, intolerable toxicity, withdrawal of informed consent, or other discontinuation criterion were met.
  Interventions: Drug: Gimistotug; Drug: BGB-15025

INTERVENTIONS:
Drug: Gimistotug — Administered intravenously
  Other Names: BGB-A445
Drug: Docetaxel — 75 milligrams per square meter (mg/m^2) administered intravenously
  Arms: Gimistotug + Docetaxel
Drug: BGB-15025 — Administered orally
  Arms: Gimistotug + BGB-15025

SUMMARY:
The main objective of this study was to evaluate the anti-tumor activity of gimistotug (BGB-A445) plus investigational agents in participants with non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study tested whether gimistotug in combination with other agents could help treat participants with non-small cell lung cancer (NSCLC) who were already treated with other anticancer agents, including anti-programmed cell death protein-1 (anti-PD-1) and anti-programmed cell death protein ligand-1 (anti-PD-L1) antibodies and platinum-based chemotherapy. The main goal of this study was to see if gimistotug could increase participant response to treatment, also called the overall response rate.

Only a portion of patients with advanced solid tumors have a durable response to currently available treatments. This represents an unmet medical need to develop improved therapeutic options. Combining immunotherapies with agents having different mechanism of action might improve outcomes for these patients.

This study was designed as a proof of concept to show that gimistotug-based combination treatment may be able to improve responses and clinical benefit in patients with NSCLC. Treatments in all cohorts was administered up to 36 cycles (approximately 2 years) until participants experienced no benefits, too many side effects, or withdrew consent.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic NSCLC (nonsquamous or squamous) that is histologically or cytologically confirmed
* Participants who have received no more than 2 lines of prior systemic therapies which must include anti-programmed cell death protein ligand-1 (anti-PD-(L)1) treatment and a platinum-based chemotherapy administered in combination with, or sequentially before or after the anti-PD-(L)1 treatment
* At least 1 measurable lesion as defined per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function as indicated by laboratory values during screening

Exclusion Criteria:

* With mixed small cell lung cancer
* Has received prior therapy targeting OX40 or any other T-cell agonists
* Has received prior therapy containing docetaxel and/or ramucirumab for advanced or metastatic NSCLC
* Has received any Chinese herbal medicine or Chinese patent medicines used to control cancer ≤ 14 days before the first dose of study drug(s)
* Active leptomeningeal disease or uncontrolled and untreated brain metastasis

NOTE: Other criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (18):
- China (15):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Hospital of Jiangnan University South Campus, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, Suwon, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Started | 21 | 14
Received Study Drug | 21 | 14
Completed | 0 | 0
Not Completed | 21 | 14
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Closed by Sponsor | 6 | 6
Not completed — Death | 12 | 7
Not completed — Declined Follow-Up Contact | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025 | Total
Number analyzed (Participants) | 21 | 14 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 11 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.48 (8.892) | 61.36 (9.532) | 62.03 (9.031)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 16 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 14 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 14 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the percentage of participants with best overall response (BOR) of a confirmed complete response (CR) or partial response (PR) as assessed by the investigators per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1.
  CR is defined as:
  * Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  * Disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes must be nonpathological in size (< 10 mm short axis).
  * No new lesions.
  PR is defined as:
  * At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * Non-progressive disease with regard to non-target lesions, persistence of 1 or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.
  * No new lesions.
Time Frame: Response was assessed every 6 weeks for the first 9 months and every 12 weeks thereafter; maximum time on follow-up was up to 13.5 months
Population: The Intent-to-Treat population included all participants who were enrolled or randomized to a treatment cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 21 | 14
percentage of participants | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 23.2]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not.
  An SAE is any untoward medical occurrence that, at any dose, meet any of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires hospitalization or prolongation of existing hospitalization
  * Results in disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is considered a significant medical AE by the investigator or the sponsor based on medical judgement
Time Frame: From first dose of study drug to 30 days after last dose. Maximum time on treatment was 11.2 months
Population: The Safety Analysis Set included all participants who were enrolled or randomized and received any dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 21 | 14
Participants
  Number of Participants Experiencing TEAEs | 20 | 12
  Number of Participants Experiencing SAEs | 8 | 1

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first determination of an objective response as assessed by the investigator per RECIST v1 until the first documentation of progression or death, whichever comes first. Median DOR was estimated using the Kaplan-Meier method.
Time Frame: From first dose to the end of study; maximum time on follow-up was up to 13.5 months.
Population: The Intent-to-Treat Analysis Set included all participants who were enrolled or randomized to a treatment cohort. Only responders were included in the analysis. No participants had a confirmed CR or PR.
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with BOR of a CR, PR, or stable disease.
  Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, with no new lesions.
Time Frame: From first dose to the end of study; maximum time on follow-up was up to 13.5 months
Population: The Intent-to-Treat Analysis Set included all participants who were enrolled or randomized to a treatment cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 21 | 14
percentage of participants | 71.4 [47.8 to 88.7] | 21.4 [4.7 to 50.8]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with BOR of a CR, PR, or stable disease lasting ≥ 24 weeks.
Time Frame: Assessed from first dose to the end of the study. Response was assessed every 6 weeks for the first 9 months and every 12 weeks thereafter; maximum time on follow-up was up to 13.5 months
Population: The Intent-to-Treat Analysis Set included all participants who were enrolled or randomized to a treatment cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 21 | 14
percentage of participants | 19.0 [5.4 to 41.9] | 0.0 [0.0 to 23.2]

6. Secondary Outcome: Serum Concentrations of Gimistotug
Time Frame: Cycle 1 Day 1 0.5 hours post-dose, Cycle 2 Day 1 predose, Cycle 5 Day 1 pre- and 0.5 hours post-dose, Cycle 9 Day 1 Predose, End of Treatment visit (30 days after last dose)
Population: The Pharmacokinetic Analysis Set included all participants who received any dose of study drug and for whom the valid study drug pharmacokinetic parameters could be estimated. Results included participants with data available at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 21 | 14
µg/mL
  Cycle 1 Day 1 Postdose 0.5 Hours | 737.95 (54) | 846.58 (18)
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 19 | 13
  Cycle 2 Day 1 Predose | 99.84 (57) | 105.90 (100)
  Cycle 5 Day 1 Predose: number analyzed (Participants) | 9 | 2
  Cycle 5 Day 1 Predose | 163.77 (113) | 222.92 (4)
  Cycle 5 Day 1 Postdose 0.5 Hours: number analyzed (Participants) | 8 | 2
  Cycle 5 Day 1 Postdose 0.5 Hours | 1027.57 (45) | 935.41 (9)
  Cycle 9 Day 1 Predose: number analyzed (Participants) | 1 | 0
  Cycle 9 Day 1 Predose | 244.00 |
  End of Treatment Visit: number analyzed (Participants) | 8 | 7
  End of Treatment Visit | 109.90 (106) | 176.79 (23)

7. Secondary Outcome: Plasma Concentrations of BGB-15025
Time Frame: Cycle 1 Day 1 2 hours and 4-6 hours post-dose, Cycle 1 Day 8 pre-dose, Cycle 1 Day 15 pre-dose, Cycle 2 Day 1 pre-dose and 2 hours and 4-6 hours post-dose, Cycle 3 Day 1 pre-dose
Population: The Pharmacokinetic Analysis Set included all participants who received any dose of study drug and for whom the valid pharmacokinetic parameters can be estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Gimistotug + BGB-15025
Number analyzed (Participants) | 14
µg/mL
  Cycle 1 Day 1 Postdose 2 Hours | 0.36 (214)
  Cycle 1 Day 1 Postdose 4-6 Hours | 0.49 (47)
  Cycle 1 Day 8 Predose | 0.29 (50)
  Cycle 1 Day 15 Predose | 0.25 (61)
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 12
  Cycle 2 Day 1 Predose | 0.18 (132)
  Cycle 2 Day 1 Postdose 2 Hours: number analyzed (Participants) | 13
  Cycle 2 Day 1 Postdose 2 Hours | 0.47 (38)
  Cycle 2 Day 1 Postdose 4-6 Hours: number analyzed (Participants) | 13
  Cycle 2 Day 1 Postdose 4-6 Hours | 0.59 (30)
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 4
  Cycle 3 Day 1 Predose | 0.30 (27)

8. Secondary Outcome: Number of Participants With Anti-Drug Antibodies to Gimistotug
Time Frame: Up to 30 days following last dose. Maximum time on treatment was 11.2 months.
Population: The Anti-Drug Antibody Analysis Set included all participants who received the study drug and in whom both baseline anti-drug antibody and at least one postbaseline anti-drug antibody results are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
Number analyzed (Participants) | 18 | 13
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 13.5 months AEs: From first dose of study drug to 30 days after last dose. Maximum time on treatment was 11.2 months
Arm/Group | Gimistotug + Docetaxel | Gimistotug + BGB-15025
All-Cause Mortality (participants affected / at risk) | 12/21 | 7/14
Serious Adverse Events (participants affected / at risk) | 8/21 | 1/14
Other Adverse Events (participants affected / at risk) | 20/21 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gimistotug + Docetaxel (N=21) | Gimistotug + BGB-15025 (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gimistotug + Docetaxel (N=21) | Gimistotug + BGB-15025 (N=14)
Anaemia (Blood and lymphatic system disorders) | 10 (14) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Asthenia (General disorders) | 5 (5) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood corticotrophin decreased (Investigations) | 1 (1) | 0 (0)
Blood corticotrophin increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Interleukin level increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (6)
Neutrophil count decreased (Investigations) | 11 (22) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 5 (10) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Anoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT06029127/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT06029127/SAP_001.pdf